CLINICAL TRIAL: NCT04572074
Title: Pilot Study to Evaluate Virtual Reality for Cancer Pain Management
Brief Title: Virtual Reality for Cancer Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Hunter Groninger, Associate Professor of Medicine, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-240
Record Dates: First submitted 2020-08-29; First posted 2020-10-01 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Cancer; Cancer Pain
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Guided imagery) (Active Comparator): 10 minutes of guided imagery experience
  Interventions: Other: Guided imagery
- Arm 2 (Virtual reality) (Experimental): 10 minutes of virtual reality experience
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Guided imagery — 10 minutes of guided imagery experience
  Arms: Arm 1 (Guided imagery)
Other: Virtual reality — 10 minutes of virtual reality experience
  Arms: Arm 2 (Virtual reality)

SUMMARY:
The purpose of this research project is to evaluate the impact of virtual reality therapy on mitigating cancer pain in hospitalized patients with cancer and compare this impact to that of 2-dimensional guided imagery distraction therapy. The purpose is also to evaluate acceptability of and satisfaction with virtual reality therapy and to examine racial and cultural preferences related to virtual reality and guided imagery thematic content.

DETAILED DESCRIPTION:
Subjects hospitalized at MedStar Washington Hospital Center will be considered for enrollment in this study if able to provide consent, at least 18 years old, and report moderate-severe pain (at least 4 out of 10 where pain is rated on a Likert scale between zero and 10) in the previous 24 hours. Subjects will be excluded if they already use VR for personal use, have intractable nausea/vomiting, history of motion sickness, history of seizures or epilepsy, have cranial structure abnormalities that prevent use of VR headset, are currently enrolled in a palliative care or pain management study, and/or are on contact isolation. Institutional review board approval will be sought and informed consent will be conducted before enrolling every patient.

After consenting to participate, in addition to usual pharmacologic pain management, 128 patients will be randomized with a 1:1 ratio to receive either one 10-minute VR session, or one 10-minute 2-dimensional guided-imagery session. The investigators believe this sample size is easily achievable given current palliative consult volumes for patients with cancer at the study institution (see above); this sample size accounts for estimates that only approximately half of eligible subjects are interested in trying VR therapies.

VR sessions will be administered using the Facebook (Facebook Inc., Menlo Park, CA) Oculus Quest VR and Touch controllers. This equipment was selected because it is portable and can be set up at the bedside in private or shared patient rooms. The hand controllers facilitate immersive, interactive VR experiences for patients who may be bedbound or have limited mobility in the inpatient setting. The VR software, Forest of Serenity (Holosphere VR ®, Birmingham, UK) is a free application that features seven non-violent mini-games in a carnival environment that can be played in a seated or fixed position.

The guided-imagery session depicts a peaceful walk through a forest with instrumental background music and 2-dimensional imagery. Subjects will watch the guided imagery video on a portable tablet for 10 minutes, the same duration as the VR intervention. Subjects in both arms will continue to receive standard pharmacologic pain management. Because of the nature of the compared interventions, subjects and researchers cannot be blinded to intervention.

The primary outcome measure will determine the impact of distraction therapy (either VR therapy or 2-dimensional guided imagery) on self-reported pain experience. Self-reported pain experience remains the standard for clinical pain research. Secondary outcomes will measure impact of each distraction therapy on general distress level, general quality of life, and satisfaction with pain management. For patients receiving opioid therapies for pain in the preceding 24 hours, the investigators will also evaluate "as needed" opioid use.

Following consent and randomization, subjects will complete surveys on electronic tablets to provide baseline data on pain scores, general distress, general quality of life, and satisfaction with pain management. Pain will be assessed using the Brief Pain Inventory-Short Form (BPI-SF, modified to assess symptoms in the last 24 hours) that includes a 0-10 Likert scale for self-reported pain as well as information about pain location, quality, and interference of pain on daily living. General distress will be measured using the Distress Thermometer (a Likert scale measuring from No Distress to Extreme Distress, where "distress" is defined by the patient). General quality of life will be measured using the Functional Assessment in Chronic Illness-Therapy in Palliative Care 14-item (FACIT-Pal 14) scale that measures non-pain symptoms and general well-being. Subjects will also be surveyed regarding comfort with technology and self-directed use of passive and active distraction therapies.

After completion of baseline surveys, subjects will be administered either VR therapy for 10 minutes or 2-dimensional guided imagery for 10 minutes. For both arms, a member of the research team will educate the subject on the technology and assure comfort with use, remaining outside the room but nearby during the actual 10 minutes.

Following the distraction therapy, subjects will be re-surveyed BPI-SF, FACIT-Pal 14, and Distress Thermometer. Both groups will also be surveyed and given semi-structured interviews regarding acceptance of and satisfaction with the distraction therapy intervention itself and its thematic content. Subjects randomized to VR therapy will be surveyed regarding level of immersion of the VR experience (Immersive Tendencies Questionnaire, http://w3.uqo.ca/cyberpsy/docs/qaires/immersion/ITQ_va.pdf).

In order to evaluate any residual effects of the distraction therapy, enrollees will be re-surveyed BPI-SF, FACIT-Pal 14, Distress Thermometer, and pain management satisfaction questions on the following day.

This study will reach 80% power to detect a difference of 1 unit in the pain score measure between the 2 groups using a two-sample t-test with equal variance at a two-sided alpha=0.05 and assuming a within-group standard deviation of 2 for each group. Sample size calculations were conducted in PASS.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized, with primary diagnosis of cancer
* age 18 and older
* report moderate-severe pain (at least 4 out of 10 where pain is rated on a Likert scale between zero and 10) in the previous 24 hours

Exclusion Criteria:

* already use VR for personal use
* intractable nausea/vomiting
* history of motion sickness
* history of seizures or epilepsy
* have cranial structure abnormalities that prevent use of VR headset
* currently enrolled in a palliative care or pain management study
* on contact isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in self-reported pain score from baseline to immediately after assigned intervention | Baseline and again immediately after assigned intervention
  Likert scale 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Change in self-reported distress from baseline to immediately after assigned intervention | Baseline and immediately after intervention, 24 hours after intervention
  National Comprehensive Cancer Network Distress Thermometer
Change in self-reported quality of life from baseline to immediately after assigned intervention | Immediately after assigned intervention
  Functional Assessment in Chronic Illness-Therapy in Palliative Care 14-item scale (FACIT Pal 14 scale) -- subject replies to 14 questions about quality of life issues with responses in 5-point Likert scale (0 = not at all; 4 = very much), total score range 0-56
Acceptability of intervention ("Would you use this intervention again?") -- this single question designed for this study | Immediately after intervention
  Single best answer: subjects choose between two choices, "Yes" or "No"
Level of immersion experienced in virtual reality arm | Immediately after intervention (virtual reality arm only)
  Immersive Experience Questionnaire
Ease of intervention ("How easy was this technology for you to use?") -- this single question designed for this study | Immediately after assigned intervention
  Single best answer to this question: subjects choose between "easy," "normal," or "difficult"
Change in self reported distress from baseline to Immediately after assigned intervention | Immediately after assigned intervention
  National Comprehensive Cancer Network Distress Thermometer -- subject rates distress at that point in time on Likert scale 0-10 (0 = no distress; 10 = worst distress)

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No